CLINICAL TRIAL: NCT03159312
Title: Influence of a Moderate Physical Exercise Program in Health of Patients Underwent Bariatric Surgery in Talca City, Chile
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, María José Aguilar Cordero, Professor, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23/01/2017 UGR
Record Dates: First submitted 2017-04-03; First posted 2017-05-18 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Bariatric Surgery Candidate
Keywords: obesity,bariatric surgery,physical activity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Assigned Interventions (Experimental): 20 individuals undergoing bariatric surgery and post surgery normal indications with moderate exercise program
  Interventions: Behavioral: Physical activity based on a moderate exercise program
- Control group (No Intervention): Control group: 23 individuals undergoing bariatric surgery and post surgery normal indications without exercise program

INTERVENTIONS:
Behavioral: Physical activity based on a moderate exercise program — Physical exercise program begins with a 2-week adaptation stage, climbs onto the treadmill (HP Cosmos®). The programming of the tape will be done initially with an intensity of 40% of its FCdRes obtained from the formula of Karvonen after performing the 6-minute walk test, you will have to maintain that intensity for 15 min, the patient is evaluated with the Borg scale and oxygen saturation permanently.After two weeks of adaptation, the HRdRes becomes to be calculated, 59% of said frequency will be modified until the exercise program is completed.The training is 30 minutes in the tradmill machine.The work of muscle strengthening of biceps, triceps, deltoids and pectorals, will be progressive in intensity and number of repetitions, determined by the evaluation of 1 Rmax. The start of work with weights is 40% of the Rmax, it will be modified monthly from 40% to 75%. Cycloergometer training (Monark ®) is without load for 15 minutes.
  Arms: Assigned Interventions

SUMMARY:
Obesity is a multifactorial disorder resulting from multivariate etiopathogenic factors. The current lifestyle, causes a gradual increase in weight both in the adult population and in the child population. Among their treatments is bariatric surgery. About which there is little evidence in the literature regarding the health condition developed by patients operated on the same. Objective: To know the influence of a moderate exercise program on health status in patients operated on with bariatric surgery. Methodology: A controlled clinical trial, the population will consist of 32 women and 11 men. Coming from the consultations of bariatric surgery of the Clinic of the Maule - Talca. In the period between March 2017 and March 2018. It will be selected following a non-probabilistic sampling and for convenience. Results Analysis: The variables used in this study will be: cardiovascular function, respiratory function, strength, health perception, anthropometric measures and functional capacity to perform exercises. The Shapiro-Wilk normality test will be performed to determine the distribution of the data to be analyzed. The t-student test or its nonparametric counterpart will be applied to compare two variables. To compare three or more variables, the ANOVA or Kruskal-Wallis test will be used depending on the results of the normality test.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Do not suffer any absolute contraindication.
* Patients who will undergo bariatric surgery and who reside in the city of Talca.
* Age between 18 - 60 years.
* With weight <180 kilograms.

Exclusion Criteria:

* Medical indication for basic pathologies.
* Post-operative complications.
* Acute angina-like pain during the 6-minute gait test.
* Absence of 2 or more trainings in a row.
* Pregnancy within the first 6 months post-surgery.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2018-03-15 (Actual); Study Completion 2018-03-18 (Actual)

PRIMARY OUTCOMES:
Quality of life prior to bariatric surgery and subsequent | 1 year
  Nottingham Scale: It is a generic instrument for measuring the physical, psychological and social suffering associated with medical, social and emotional problems of the extent to which such suffering affects the lives of individuals, and ICIQ-SF urinary incontinence questionnaire

SECONDARY OUTCOMES:
Blood sugar level | 1 year
  Hemoglucotest, for measuring peripheral blood glucose
Quality of sleep | 1 year
  Pittsburgh Sleep Quality Questionnaire
Anthropometric measures | 1 year
  Rosscraft anthropometry kit containing Campbell 20 (Campbell 10) and Bioelectrical impedance.
Level of physical ability | 1 year
  Borg scale
Level of physical ability | 1 year
  6-minute walk test
Perception of health | 1 year
  Assessment pre-operated patients bariatric surgery
Cardiovascular function | 1 year
  With dynamometer
Cardiovascular function | 1 year
  Tensiometers cable
Cardiovascular function | 1 year
  Cells of load.
Strength | 1 year
  To analyze the strength and the dynamic resistance were used: free weights (dumbells and bars) exercise machines with constant, variable or isokinetic resistance

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Granada, Granada, Spain